CLINICAL TRIAL: NCT05851612
Title: Comparison of PEEP Titration Guided by Driving Pressure Versus Oxygenation Method Versus Constant PEEP in Patients Undergoing Esophagectomy With One Lung Ventilation in Prone Position
Brief Title: Comparison of Three Methods of PEEP Titration During One Lung Ventilation in Prone Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amany Hazem abdelmaksood EL-deeb, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEEP in OLV in prone position
Record Dates: First submitted 2023-04-14; First posted 2023-05-09 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: One Lung Ventilation
Keywords: optimal PEEP -one lung ventilation-prone position

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: A single investigator will assess the patients for eligibility, obtain written informed consent, open the sealed opaque envelopes containing group allocation and set up the ventilator as specified in the envelope. The study subjects and the resident assessing the outcome will be blinded to the study group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group C(constant group) (Active Comparator): Constant PEEP of 5 centimeter of water (cm H2O) will be applied
  Interventions: Procedure: constant PEEP
- group D (driving group) (Active Comparator): PEEP titration will be according to driving pressure
  Interventions: Procedure: Driving pressure guided PEEP
- group O (oxygenation group) (Active Comparator): PEEP titration will be according to oxygenation method
  Interventions: Procedure: oxygenation method guided PEEP

INTERVENTIONS:
Procedure: constant PEEP — Constant PEEP of 5 cm H2O will be applied and maintained throughout one-lung ventilation.
  Arms: group C(constant group)
Procedure: Driving pressure guided PEEP — PEEP titration will be started at 5 cmH2O and then increased in 1 cmH2O interval to 10 cmH2O. After 10 breath cycles will maintained, Driving pressure (ΔP) will be measured at each PEEP level at the last cycle. The PEEP indicating the lowest ΔP will be selected if multiple levels of PEEP showed the same lowest ΔP, the lowest PEEP will be selected. Driving pressure will be calculated as plateau pressure minus PEEP. Titration will stopped if peak inspiratory pressure of 50 cm H2O, or plateau pressure of 40 cm H2O reached, or hypotension will be observed.
  Arms: group D (driving group)
Procedure: oxygenation method guided PEEP — PEEP titration will be started from 5 cmH2O and increase of 1 cmH2O every 4 min with fixed driving pressure that will result in delivery of a fixed tidal volume (TV) of 6ml/kg ideal body weight (IBW). Optimal PEEP will be defined as the PEEP below which PaO2 /FIO2 falls by at least 20%. If at least 20% PaO2 /FIO2 decrement is not obtained, then PEEP that will result in the highest PaO2 will be selected.
  Arms: group O (oxygenation group)

SUMMARY:
One-lung ventilation and prone positioning during thoracoscopic esophagectomy is associated with pulmonary complications so lung protection is strongly recommended. Individualization the optimal PEEP level according to the respira¬tory condition of patients has gradually attracted the attention of clinicians. The aim of this study is to compare and evaluate the differences between three different PEEP values in patients who will undergo thoracoscopic esophagectomy receiving either constant PEEP or driving pressure guided individualized PEEP or oxygenation guided individualized PEEP.

DETAILED DESCRIPTION:
Induction of general anesthesia and mechanical ventilation impair respiratory function because of alveoli collapse, decreased functional residual capacity, diminished arterial oxygenation, and even mechanical ventilation-induced injury.In addition, One-lung ventilation during thoracic surgery is prone to ventilator induced lung injury and oxygen toxicity. It is also associated with a profound inflammatory cytokine release which causes excessive neutrophils recruitment that increases pulmonary vascular permeability in both lungs. These reactions often precede systemic inflammatory response syndrome, acute respiratory distress syndrome and pneumonia. Therefore, lung protection and protective ventilation is strongly recommended during thoracic surgery.In contrast to the lateral decubitus position, OLV in the prone position is devoid of the beneficial effect of gravity on preferential redistribution of the pulmonary blood flow to the dependent areas of a lung, possibly resulting in increased V/Q mismatch. Also, the prone position is frequently associated with decreased respiratory compliance and increased peak airway pressure in anesthetized and paralyzed patients when not assuring free abdominal and chest movements, which is further aggravated by CO2 insufflation. Prone positioning during esophagectomy provides several advantages, including shortened operative times and superior surgical view, at the cost of one-lung ventilation (OLV). Intraoperative lung protective ventilation strategy, which includes the combination of low tidal volume and adequate PEEP levels during operation, has been reported to improve respiratory mechanics and reduce the incidence and severity of atelectasis which may prolong hospital stays and increase mortality in surgical patients.Improper PEEP levels have an impact on patient physiology. If the setting level is too low to achieve the desired purpose, it cannot produce the effect of applying PEEP. If the setting level is too high, the pulmonary vascular resistance increases, venous return blood volume decreases, intrapulmonary shunt increases, and arterial oxygen partial pressure level is reduced. Also, it could negatively affect cardiac output and delivery of oxygen to vital organs.Individualization the optimal PEEP level according to the respira¬tory condition of patients has gradually attracted the attention of clinicians. The methods to determine the best PEEP levels include computed tomography scanning, electri¬cal impedance tomography, ultrasound, P-V curve method, best oxygenation titration method, and best lung compliance titration method. Each method has its advantages and disadvantages. Individualized PEEP has advantages over fixed PEEP in improved respiratory mechanics and prevent progressive alveolar collapse.There are few studies on the selection of appropriate PEEP values during one-lung ven¬tilation (OLV) in prone position and the protective effect of PEEP values can be titrated by different titration methods which still requires many prospective studies. Therefore, this study will be conducted to compare PEEP titration using driving pressure versus oxygenation method versus constant PEEP and evaluate their efficacy on oxygenation, ventilation, hemodynamics and PPC for patients undergoing thoracoscopic esophagectomy treated with one lung ventilation in prone position.

Aim of the Study:

The aim of this study is to compare and evaluate the differences between three different PEEP values in patients who will undergo thoracoscopic esophagectomy treated with one lung ventilation in prone position receiving either constant PEEP or driving pressure guided individualized PEEP or oxygenation guided individualized PEEP.

It is hypothesized that the individualized PEEP guided by driving pressure could improve intraoperative oxygenation function, pulmonary mechanics, early postoperative atelectasis, and reduce the incidence of postoperative pulmonary complications(PPCs) for patients undergoing thoracoscopic esophagectomy treated with one lung ventilation in prone position.

Sample Size Calculation:

A pilot study was performed to measure the lung ultrasound score at the end of the surgery to estimate the sample size. Sample size calculations were performed using G. power software (version 3.1.9.7). The means and standard deviations for the D group, O group, and C group were 10.5 + 2.02, 11.7 + 1.2, and 12.5 + 2.5, respectively. Sample size calculations showed that 11 subjects per group will be required to achieve 95% power with a Type I error of 0.05. A total of 42 patients (14 patients per group) will be included in this trial considering an 80% adherence rate.

Methods:

The study will include 42 patients who will be scheduled for thoracoscopic esophagectomy treated with one lung ventilation in prone position under general anesthesia. It will be conducted in Mansoura gastroenterology center over one year and patients will be recruited in june 2023. they will be randomly assigned to 3 equal groups (D group, O group and C group) according to computer-generated table of random numbers using the permuted block randomization method. The group allocation will be concealed in sequentially numbered, sealed opaque envelopes which will be opened only after obtaining the written informed consent.A single investigator will assess the patients for eligibility, obtain written informed consent, open the sealed opaque envelopes containing group allocation and set up the ventilator as specified in the envelope. The study subjects and the resident assessing the outcome will be blinded to the study group.The study protocol will be explained to all patients after enrollment into the study. They will be kept fasting according to pre-operative ASA recommendations prior to surgery. Basic demographic characters including age, sex, and BMI will be recorded. The peri-operative management will be identical in the three groups.

Statistical analysis:- The collected data will be coded, processed, and analyzed using Statistical Package for the Social Sciences (SPSS) program (version 22) for Windows. Normality of numerical data distribution will be tested by Kolmogorov-Smirnov test. Normally distributed numerical data will be presented as mean and standard deviation, and their comparison in different groups will be performed using one-way ANOVA with post-hoc Bonferroni test. Non-normally distributed numerical data will be presented as median and range, and compared nonparametrically using Kruskal-Wallis test followed by Mann-Whitney U test. Categorical data will be presented as number and percentage, and their comparison will be performed using Chi-square test. The all data will be considered significant if P value is ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) (grade 1or 2) patients.
* Scheduled for elective thoracoscopic esophagectomy treated with one lung ventilation in prone position and surgery of expected duration greater than 1 h.
* Body mass index (BMI) less than 30 kg/m2.

Exclusion Criteria:

* Patient's refusal.
* Altered mental status or un-cooperative patients.
* History of known sensitivity to the used anesthetics.
* Significant cardiac dysfunction, hepatic, or renal impairment.
* History of severe chronic obstructive pulmonary disease.
* History of severe or uncontrolled bronchial asthma.
* History of severe restrictive lung disease.
* History of pulmonary metastases.
* History of any thoracic surgery.
* Need for chest drainage prior to surgery.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
lung ultrasound score | Up to 5 min before leaving the post anesthesia care unit (PACU)
  Thorax will be divided into 12 segments. The lung ultrasound score is 0 to 3, based on the B-line count and the degree of subpleural solidity. A total score of 0-36 will be obtained by summing the scores of the 12 segments. The absolute difference in the three lung ultrasound scores measured before induction, before neuromuscular block reversal, at the end of surgery/before extubation, and 5 min before leaving the PACU respectively.

SECONDARY OUTCOMES:
Positive end-expiratory pressure (PEEP) | Up to the end of the procedure
  It will be collected at 10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
The ratio of partial pressure of oxygen in arterial blood to the fraction of inspiratory oxygen concentration (PaO2/FiO2 ratio) | Up to the end of the procedure
  It will be collected at before induction ,10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
Heart rate (HR) | Up to the end of the procedure
  It will be recorded before the procedure, after 15 min, 30 minutes and then every 30min intraoperative till the end of surgery.
The Central venous pressure (CVP) values | Up to the end of the procedure
  It will be recorded before the procedure, after 15 min, 30 minutes and then every 30min intraoperative till the end of surgery.
The total volume of fluids and vasopressors administered | Up to the end of the procedure
  They will be recorded at the end of surgery
The duration of operation, anesthesia and one lung ventilation . | Up to the end of the procedure
  will be recorded at the end of surgery
Occurrence of Intra-operative adverse effects | Up to the end of the procedure
  Any adverse events occur intraoperative as hypotension or bradycardia will be recorded.
Plateau pressure | Up to the end of the procedure
  It will be collected at 10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
Driving pressure | Up to the end of the procedure
  It will be collected at 10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
Tidal volume | Up to the end of the procedure
  It will be collected at 10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
Static compliance | Up to the end of the procedure
  It will be collected at 10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
Peak pressure | Up to the end of the procedure
  It will be collected at 10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
End-tidal carbon dioxide | Up to the end of the procedure
  It will be collected at 10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
Oxygen saturation | Up to the end of the procedure
  It will be collected at 10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
The alveolar-arterial gradient (A-a gradient) | Up to the end of the procedure
  It will be collected at 10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
the potential of hydrogen (pH) | Up to the end of the procedure
  It will be collected at before induction ,10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
The partial pressure of carbon dioxide in arterial blood(PaCO2) | Up to the end of the procedure
  It will be collected at before induction ,10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
the partial pressure of oxygen n arterial blood(PaO2) | Up to the end of the procedure
  It will be collected at before induction ,10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
Actual base excess | Up to the end of the procedure
  It will be collected at before induction ,10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
Bicarbonate (HCO3) | Up to the end of the procedure
  It will be collected at before induction ,10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
Lactate | Up to the end of the procedure
  It will be collected at before induction ,10 minutes after induction, Prone position, 10 minutes after titration and every hour until the end of OLV, before neuromuscular block reversal and at the end of surgery/before extubation.
Mean arterial blood pressure (MAP) | Up to the end of the procedure
  It will be recorded before the procedure, after 15 min, 30 minutes and then every 30min intraoperative till the end of surgery.
Occurrence of post-operative complications. | up to one week after the procedure
  the occurrence of PPC (cough, increased sputum, dyspnea, chest pain, temperature above 38 °C, HR > 100 beats/min) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Amany EL-Deeb, MD, Principal Investigator — Faculty of Medicine, Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Result] Choi YS, Shim JK, Na S, Hong SB, Hong YW, Oh YJ. Pressure-controlled versus volume-controlled ventilation during one-lung ventilation in the prone position for robot-assisted esophagectomy. Surg Endosc. 2009 Oct;23(10):2286-91. doi: 10.1007/s00464-008-0310-5. Epub 2009 Jan 30. PMID 19184209
- [Result] Wang ZY, Ye SS, Fan Y, Shi CY, Wu HF, Miao CH, Zhou D. Individualized positive end-expiratory pressure with and without recruitment maneuvers in obese patients during bariatric surgery. Kaohsiung J Med Sci. 2022 Sep;38(9):858-868. doi: 10.1002/kjm2.12576. Epub 2022 Jul 22. PMID 35866347
- [Result] Park M, Ahn HJ, Kim JA, Yang M, Heo BY, Choi JW, Kim YR, Lee SH, Jeong H, Choi SJ, Song IS. Driving Pressure during Thoracic Surgery: A Randomized Clinical Trial. Anesthesiology. 2019 Mar;130(3):385-393. doi: 10.1097/ALN.0000000000002600. PMID 30664548
- [Result] Yao W, Yang B, Wang W, Han Q, Liu F, Shan S, Wang C, Zheng M. Effect of Positive End-Expiratory Pressure (PEEP) Titration in Elderly Patients Undergoing Lobectomy. Med Sci Monit. 2022 Dec 13;28:e938225. doi: 10.12659/MSM.938225. PMID 36510453
- [Result] Liu K, Huang C, Xu M, Wu J, Frerichs I, Moeller K, Zhao Z. PEEP guided by electrical impedance tomography during one-lung ventilation in elderly patients undergoing thoracoscopic surgery. Ann Transl Med. 2019 Dec;7(23):757. doi: 10.21037/atm.2019.11.95. PMID 32042773
- [Result] Monastesse A, Girard F, Massicotte N, Chartrand-Lefebvre C, Girard M. Lung Ultrasonography for the Assessment of Perioperative Atelectasis: A Pilot Feasibility Study. Anesth Analg. 2017 Feb;124(2):494-504. doi: 10.1213/ANE.0000000000001603. PMID 27669555
- [Result] Xu Q, Guo X, Liu J, Li SX, Ma HR, Wang FX, Lin JY. Effects of dynamic individualized PEEP guided by driving pressure in laparoscopic surgery on postoperative atelectasis in elderly patients: a prospective randomized controlled trial. BMC Anesthesiol. 2022 Mar 16;22(1):72. doi: 10.1186/s12871-022-01613-9. PMID 35296253